CLINICAL TRIAL: NCT06478641
Title: Expanded Access Protocol: Use of Tafenoquine for Treatment of Babesiosis in Immunocompromised Patients With Persistent Babesia Microti Despite Prior Treatment
Brief Title: Expanded Use in Persistent (B. Microti) Babesiosis
Status: Available | Type: Expanded Access
Sponsor: 60 Degrees Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: TQ-BA-2024-2
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Persistent Babesiosis
MeSH Terms: interventions — tafenoquine

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine will be self-administered orally as 2 x 100 mg dark pink coated tablets once daily (total daily dose 200 mg) with food on Days 1, 2, 3 & 4 then weekly thereafter (starting on day 11) until the patient has two consecutive negative PCR tests for Babesia parasites and symptoms of babesiosis have resolved.

SUMMARY:
The purpose of this expanded access protocol is to offer a potentially effective treatment (tafenoquine) to patients with persistent babesiosis, who have not responded to standard of care treatments, and who are immunocompromised and thus at risk for more serious complications. Tafenoquine will be self-administered orally as 2 x 100 mg dark pink coated tablets once daily (total daily dose 200 mg) with food on Days 1, 2, 3 & 4 then weekly thereafter (starting on day 11) until the patient has two consecutive negative PCR tests for Babesia parasites and symptoms of babesiosis have resolved. Other standard of care treatments recommended in the 2020 IDSA Guideline on Diagnosis and Management of Babesiosis should also be included in the treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years
* Laboratory confirmed infection with B. microti and exhibiting clinical symptoms of babesiosis
* Able and willing to give written informed consent
* Able to take ARAKODA according to Prescribing Information
* If female willing to take birth control for 90 days
* Have risk factors for relapsing disease
* Azithromycin, atovaquone, and/or clindamycin administered in the last 12 months to treat babesiosis, and, in the opinion of the investigator, high likelihood that current infection represents a relapse or continuation of disease
* Willing to initiate or continue a standard of care antimicrobial regimen

Exclusion Criteria:

* Have any of the contraindications for ARAKODA
* Current or planned treatment with quinine while participating in the study
* Any concomitant significant illness unrelated to babesiosis
* Taking any excluded concomitant medication
* The patient is unable to tolerate medication by the oral route

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult